CLINICAL TRIAL: NCT00847106
Title: Augmentation of Dendritic Cell Based Vaccines in Melanoma Patients by Depletion of Regulatory T Cells With an Anti-CD25 Monoclonal Antibody (Daclizumab). A Clinical Study.
Brief Title: Augmentation of Dendritic Cell-Based Vaccines in Melanoma Patients by Depletion of Regulatory T Cells in Stage IV Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-2893; KWF 2003-2893
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Melanoma
Keywords: Dendritic Cells; Regulatory T cells; CD25; Melanoma; Immunotherapy; Daclizumab; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab
Biological: Dendritic cells

SUMMARY:
Dendritic cells (DC) are the professional antigen presenting cells of the immune system. Multiple distinct DC lineage's exist and it is now well appreciated that the DC subset and the maturation stage of the DC determines the type of immune response, ranging from a TH1 or TH2 response to immune tolerance. The extremely potent capacity of mature DC to initiate immune responses can be exploited to fight infectious diseases and cancer. Others and we are currently using tumor antigen loaded mature DC in clinical vaccination studies against cancer, and clinical as well as immunological responses have been observed.

Exciting new insights accompany the revival of suppressor T cells, now referred to as regulatory T cells (Treg), and implicate that also Treg play a key role in the control of immunity. Treg constitute a sub-population of CD4+ T cells constitutively expressing the IL-2R alpha-chain (CD25). Treg show remarkably suppressive activities on different components of the immune system, including T lymphocytes and dendritic cells, suggesting they act both at the initiation phase (DC) and at the effector phase (activated T cells) of the immune response. Interestingly, temporal depletion of Treg has been shown to enhance anti-tumor immune responses and in case of prolonged absence of Treg even autoimmunity. Furthermore, data in mouse tumor models indicate that temporal depletion of Treg also results in improved vaccine efficiency in the therapeutic setting, e.g. in mice with a pre-existing tumor. These data imply that in tumor bearing patients depletion of Treg prior to vaccination will improve vaccine efficacy.

In this study we investigate the effect of regulatory T cell (Treg) depletion on the efficacy of DC-based anti-tumor vaccines in a clinical study using melanoma associated antigens tyrosinase and gp100-loaded DC and a depleting anti-CD25 mononuclear antibody (Daclizumab). Our primary objective in this study is the induction of an effective anti-tumor immune response. Our secondary objective is the induction of a clinical response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented evidence of melanoma.
2. Stage IV melanoma according to the 2001 AJCC criteria. [53] Limited tumor burden; LDH < 2x upper limit of normal.
3. HLA-A2.1 phenotype according to lymphocyte HLA typing.
4. Expression of gp100 and/or tyrosinase on melanoma cells, as detected by immunohistochemistry, preferably on metastatic tumor, but if not available on primary tumor.
5. ECOG performance status 0-1, life expectancy > 3 months.
6. Age 18-75 years. -
7. Written informed consent.
8. Expected adequacy of follow-up.
9. WBC > 3.0 x 109/l, lymphocytes > 0.8 x 109/l, platelets > 100 x 109/l, serum creatinine < 150 μmol/l, serum bilirubin < 25 μmol/l.

   Exclusion Criteria:
10. No clinical signs of CNS metastases, in patients with a clinical suspicion of CNS metastases CT scan of the brain should be performed to exclude this.
11. No prior chemotherapy, immunotherapy, or radiotherapy within three months before planned vaccination is allowed.
12. No previous treatment with monoclonal antibodies.
13. No concomitant use of corticosteroids or other immunosuppressive agents.
14. No history of second malignancy within the last 5 years. Adequately treated basal carcinoma of skin or carcinoma in situ of cervix is acceptable within this period.
15. No serious concomitant disease, no active infections. Specifically, patients with autoimmune disease or organ allografts, and HBsAg or HIV positive patients are excluded.
16. Patients with a known allergy to shell fish (contains KLH) are excluded.
17. Patients with asthma or severe allergic disease necessitating medication are excluded
18. No pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10

PRIMARY OUTCOMES:
Immune reponse

SECONDARY OUTCOMES:
Clinical Response

CONTACTS AND LOCATIONS:
Overall Officials: Prof. C.J.A. Punt, MD, PhD, Principal Investigator — Radboud University Medical Center; Prof. G.J. Adema, PhD, Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Background] Sutmuller RP, van Duivenvoorde LM, van Elsas A, Schumacher TN, Wildenberg ME, Allison JP, Toes RE, Offringa R, Melief CJ. Synergism of cytotoxic T lymphocyte-associated antigen 4 blockade and depletion of CD25(+) regulatory T cells in antitumor therapy reveals alternative pathways for suppression of autoreactive cytotoxic T lymphocyte responses. J Exp Med. 2001 Sep 17;194(6):823-32. doi: 10.1084/jem.194.6.823. PMID 11560997
- [Background] de Vries IJ, Bernsen MR, Lesterhuis WJ, Scharenborg NM, Strijk SP, Gerritsen MJ, Ruiter DJ, Figdor CG, Punt CJ, Adema GJ. Immunomonitoring tumor-specific T cells in delayed-type hypersensitivity skin biopsies after dendritic cell vaccination correlates with clinical outcome. J Clin Oncol. 2005 Aug 20;23(24):5779-87. doi: 10.1200/JCO.2005.06.478. PMID 16110035
- [Background] De Vries IJ, Krooshoop DJ, Scharenborg NM, Lesterhuis WJ, Diepstra JH, Van Muijen GN, Strijk SP, Ruers TJ, Boerman OC, Oyen WJ, Adema GJ, Punt CJ, Figdor CG. Effective migration of antigen-pulsed dendritic cells to lymph nodes in melanoma patients is determined by their maturation state. Cancer Res. 2003 Jan 1;63(1):12-7. PMID 12517769
- [Background] Lesterhuis WJ, de Vries IJ, Adema GJ, Punt CJ. Dendritic cell-based vaccines in cancer immunotherapy: an update on clinical and immunological results. Ann Oncol. 2004;15 Suppl 4:iv145-51. doi: 10.1093/annonc/mdh919. No abstract available. PMID 15477299
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] de Vries IJ, Lesterhuis WJ, Scharenborg NM, Engelen LP, Ruiter DJ, Gerritsen MJ, Croockewit S, Britten CM, Torensma R, Adema GJ, Figdor CG, Punt CJ. Maturation of dendritic cells is a prerequisite for inducing immune responses in advanced melanoma patients. Clin Cancer Res. 2003 Nov 1;9(14):5091-100. PMID 14613986
- [Background] de Vries IJ, Eggert AA, Scharenborg NM, Vissers JL, Lesterhuis WJ, Boerman OC, Punt CJ, Adema GJ, Figdor CG. Phenotypical and functional characterization of clinical grade dendritic cells. J Immunother. 2002 Sep-Oct;25(5):429-38. doi: 10.1097/00002371-200209000-00007. PMID 12218781
- [Background] Adema GJ, de Vries IJ, Punt CJ, Figdor CG. Migration of dendritic cell based cancer vaccines: in vivo veritas? Curr Opin Immunol. 2005 Apr;17(2):170-4. doi: 10.1016/j.coi.2005.01.004. PMID 15766677
- See also: website of the Radboud University Nijmegen Medical Centre — http://www.umcn.nl